CLINICAL TRIAL: NCT04340765
Title: Comparative Evaluation of Metastatic Lesions From Prostate Carcinoma With 18F-NaF and 18F-Fluorocholine PET/CT
Brief Title: 18F-fluorocholine and 18F-fluoride PET in Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB106-65-A
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Prostate Cancer; Fluorocholine
Keywords: Prostate cancer; NaF; Bone scan; 18F-Fluorocholine; PET
MeSH Terms: conditions — Prostatic Neoplasms | interventions — fluorocholine

STUDY DESIGN:
Intervention Model Description: The patients will receive both 18F-fluorocholine PET and NaF PET
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 18F-fluorocholine PET/CT (Experimental): 18F-fluorocholine PET/CT
  Interventions: Drug: 18F-fluorocholine

INTERVENTIONS:
Drug: 18F-fluorocholine — Dual phase 18F-fluorocholine PET/CT
  Other Names: 18F-NaF

SUMMARY:
Prostate cancer remains to be a public health problem around the world. For patients with prostate cancer, diphosphonate bone scintigraphy (BS) and pelvic tomographic imaging are major imaging tools to evaluate the disease spread. However, the conventional image modalities have only limited sensitivity and specificity. New imaging tracer with 18F-fluorocholine (18F-FCH) and old radiopharmaceuticals with NaF has showed promising results in detecting prostate cancers over bone scan. Nevertheless, the diagnostic performance of each tool has less been compared.

The goal of this study is to compare the diagnostic performance of 18F-FCH PET/CT and NaF PET/CT for prostate cancer patients.

The investigators prospectively enroll patients with the pathological diagnosis of prostate cancer and intended to receive radionuclide bone image. The patients will receive NaF PET/CT and 18F-FCH PET/CT. Each image will be evaluated by experienced interpreter for abnormal uptake suspicious for cancer spreading. The reference standard will be a combination of tissue correlation, imaging, laboratory and clinical data. Diagnostic performance of both PET/CT scans will be measured and calculated.

DETAILED DESCRIPTION:
The investigators conducted a prospective study to investigate the performance of 18F-choline (FCH) PET/CT and 18F-NaF PET in the patients with prostate adenocarcinoma.

18F-NaF PET imaging protocol: Fasting is not needed before radiotracer injection. No specific drug restriction is needed. Scan will be conduced by using a PET/CT unit (Discovery ST; GE Medical Systems, Milwaukee,Wis), and scans will be interpreted on a work station with the use of compatible software (Xeleris).

An indwelling intravenous catheter connected to an infusion line and an saline syringe will be set on each patient. 18F-NaF (148 +/- 10% MBq) will be injected intravenously through the infusion line and will be flushed by saline. NaF PET/CT scan acquisition is to be taken 30 minutes after radiotracer injection. The PET/CT (120 mA, 120 kVp) scan field will cover from vertex to toe.

Image analysis: Two nuclear medicine physicians assess the NaF PET/CT images. The investigators have access to the patients' history and interpreted individually by each reader, with disagreements to be resolved by consensus. Uptake in the focus will be evaluated of the likelihood of cancer in 5-graded scale. 0. No cancer or definitely no pathologic aspect; 1. Probably benign lesion; 2. Equivocal lesion; 3. Probably cancer; 4. Most probably cancer. For the determination of a diagnosis, score 0 and 1 are considered a negative result and 2 to 4 a positive result.

18F-FCH PET imaging protocol: The 18F-FCH PET will be arranged within 6 weeks after NaF PET. Fasting is not needed before radiotracer injection. No specific drug restriction is needed. Scan will be conduced by using a PET/CT unit (Discovery ST; GE Medical Systems, Milwaukee,Wis), and scans will be interpreted on a work station with the use of compatible software (Xeleris).

An indwelling intravenous catheter connected to an infusion line and an saline syringe will be set on each patient. 18F-FCH (185 +/- 10% MBq) will be injected intravenously through the infusion line and will be flushed by saline. The injected 18F-FCH dose, injection time, post-injection residual activity, time of start imaging and time of end imaging will be recorded on case report form. 18F-FCH PET/CT scan acquisition is to be taken 5 to 10 minutes after radiotracer injection. The PET/CT (80-120 mA, 120 kVp) scan field will cover from skull to mid-thigh. The 18F-FCH PET/CT scan time will require 35-40 minutes.

Image analysis: Two nuclear medicine physicians assess the 18F-FCH PET/CT images. The investigators have access to the patients' history and interpreted individually by each reader, with disagreements to be resolved by consensus. Uptake in the focus will be evaluated of the likelihood of cancer in 5-graded scale. 0. No cancer or definitely no pathologic aspect; 1. Probably benign lesion; 2. Equivocal lesion; 3. Probably cancer; 4. Most probably cancer. For the determination of a diagnosis, score 0 and 1 are considered a negative result and 2 to 4 a positive result.

Reference standard: The skeletal lesion will be evaluated by both 18F-FCH PET/CT and NaF PET/CT findings. Congruent positive lesion and congruent negative will be defined as true positive and true negative, respectively. A third image study (MRI or CT) will be introduced for those with incongruent and ambiguous PET features. Biopsy will be reserved for those lesions with undetermined results after third image study.

The extra-skeletal cancerous lesions are theoretically be detected on 18F-FCH PET/CT only, thus, the reference modality will not include NaF PET/CT. The prostate bed in patients with either positive or negative imaging studies will be investigated with pelvic MRI. Patients with abnormal foci in pelvic and abdominal extraprostatic tissue at imaging will be investigated by using pelvic MRI as well. If lesions on MRI and 18F-FCH PET/CT are both positive, the lesions will be treated as malignancy. Patients with lesions on 18F-FCH PET/CT along will be evaluated by the investigator and co-investigators to decide if the patient will receive biopsy or not. The lesion will be confirmed to be malignant if positive biopsy results. The patient will receive further follow-up by MRI and serum PSA after 6 and 12 months if the patient is not suitable for biopsy. The lesion will be confirmed to be malignant if substantial growth in lesion size or increase serum PSA. Patients with both negative MRI and negative 18F-FCH PET/CT will be evaluated by the aforementioned follow-up schedule as well. If the initial pelvic MRI is positive for malignancy and the 18F-FCH PET/CT is negative, the lesion will be treated as positive for malignancy. However, the patient still need the 6 and 12 months of follow-up to confirm the nature of the lesion. Biopsy will be reserved for those patients with undetermined results despite vigorous image studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients are pathologically diagnosed with prostate adenocarcinoma.
* Received NaF PET/CT.

Exclusion Criteria:

* Diagnosed to have multiple cancers
* Younger than 20-year-old
* Known allergic to investigational drug
* The patients is classified as not suited for the exam by the investigators.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The sensitivities of 18F-fluorocholine PET/CT and NaF PET/CT | 6 weeks
  The lesion-based sensitivities of these two image modalities (The number of true positive image findings/The number of confirmed metastasis)
The specificities of 18F-fluorocholine PET/CT and NaF PET/CT | 6 weeks
  The lesion-based specificities of these two image modalities (The number of true negative image findings/The number of confirmed e benign lesion)

SECONDARY OUTCOMES:
Extraskeletal metastatic lesions detected by 18F-fluorocholine PET/CT | 6 weeks
  To calculated the extraskeletal metastatic lesion that is detected by 18F-fluorocholine PET/CT

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hung Chen, M.D., Principal Investigator — Hualien Tzu Chi General Hospital
Locations (1):
- Hualien Tzu Chi Hospital, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No